CLINICAL TRIAL: NCT01915940
Title: A Phase 2, Multicenter, Randomized, Subject- and Examiner-masked, Controlled Clinical Trial Designed to Evaluate the Safety and Effectiveness of the Bimatoprost Ocular Insert as Compared to Topical Timolol Solution (0.5%) in Patients With Glaucoma or Ocular Hypertension.
Brief Title: Bimatoprost Ocular Insert Compared to Topical Timolol Solution in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ForSight Vision5, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FSV5-002
Record Dates: First submitted 2013-07-31; First posted 2013-08-05 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Primary Open-Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Primary Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Bimatoprost; Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 13 mg Bimatoprost Ocular Insert (Experimental): Washout and placebo ocular insert in each eye for at least 4 weeks, followed by 13 mg Bimatoprost Ocular Insert in each eye and placebo eye drops twice a day in each eye for 6 months.
  Interventions: Drug: Bimatoprost; Drug: Placebo Eye Drops; Device: Placebo Ocular Insert
- Timolol 0.5% + Placebo Ocular Insert (Active Comparator): Washout and placebo ocular insert in each eye for at least 4 weeks, followed by Timolol (timoptic ophthalmic solution 0.5%) twice a day in each eye plus placebo ocular insert for 6 months.
  Interventions: Drug: Timolol 0.5%; Device: Placebo Ocular Insert

INTERVENTIONS:
Drug: Bimatoprost — Bimatoprost ocular insert
  Arms: 13 mg Bimatoprost Ocular Insert
Drug: Timolol 0.5% — Timolol 0.5% solution
  Other Names: timoptic
  Arms: Timolol 0.5% + Placebo Ocular Insert
Drug: Placebo Eye Drops — Placebo topical eye drops
  Arms: 13 mg Bimatoprost Ocular Insert
Device: Placebo Ocular Insert — Ocular insert without any active drug
  Other Names: non-medicated (placebo) Ocular Insert

SUMMARY:
The objective of this Phase 2 study is to evaluate whether the Bimatoprost Ocular Insert is non-inferior to that of timolol ophthalmic solution (0.5%) at 12 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent
* Primary open-angle glaucoma or ocular hypertension in both eyes
* Best-corrected distance vision of 20/80 or better
* Stable visual field
* corneal thickness between 490-620 micrometers

Key Exclusion Criteria:

* Cup-to-disc ratio greater than 0.8
* significant risk of angle closure due to pupil dilation, defined as a Shaffer classification of less than grade 2 based on gonioscopy
* laser surgery for glaucoma/ocular hypertension on one or both eyes within the last 12 months
* past history of corneal refractive surgery
* past history of any incisional surgery for glaucoma at any time
* corneal abnormalities that would interfere with tonometry readings
* current participation in an investigational drug or device study or participation in such a study within 30 days of screening
* Inability to accurately evaluate the retina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2013-10-23 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Chen, PhD, Study Director — Allergan
Locations (10):
- United States (10):
  - Sall Medical Research Center, Artesia, California
  - Scripps Clinic Torrey Pines, La Jolla, California
  - Eye Research Foundation, Newport Beach, California
  - UC Davis Dept of Ophthalmology & Vision Science, Sacramento, California
  - Coastal Research Associates, Atlanta, Georgia
  - Clayton Eye Center, Morrow, Georgia
  - Ophthalmology Consultants, St Louis, Missouri
  - UNC Kittner Eye Center, Chapel Hill, North Carolina
  - Apex Eye, Madeira, Ohio
  - Ophthalmology Associates PC, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belamkar A, Harris A, Zukerman R, Siesky B, Oddone F, Verticchio Vercellin A, Ciulla TA. Sustained release glaucoma therapies: Novel modalities for overcoming key treatment barriers associated with topical medications. Ann Med. 2022 Dec;54(1):343-358. doi: 10.1080/07853890.2021.1955146. PMID 35076329

RESULTS

PARTICIPANT FLOW:
Groups:
- Washout + Placebo Ocular Insert: Glaucoma medication washout and placebo ocular insert in each eye for at least 4 weeks.
- 13 mg Bimatoprost Ocular Insert: Following the washout period, 13 mg Bimatoprost Ocular Insert and placebo eye drops twice a day in each eye for 6 months.
- Timolol 0.5% + Placebo Ocular Insert: Following the washout period, timolol ophthalmic solution 0.5% twice a day plus placebo ocular insert in each eye for 6 months.
Period: Pre-randomization Washout Period
Arm/Group | Washout + Placebo Ocular Insert | 13 mg Bimatoprost Ocular Insert | Timolol 0.5% + Placebo Ocular Insert
Started | 169 | 0 | 0
Completed | 130 | 0 | 0
Not Completed | 39 | 0 | 0
Not completed — Not Qualified for Randomization | 39 | 0 | 0
Period: Treatment Period
Arm/Group | Washout + Placebo Ocular Insert | 13 mg Bimatoprost Ocular Insert | Timolol 0.5% + Placebo Ocular Insert
Started | 0 | 64 | 66
Completed | 0 | 53 | 62
Not Completed | 0 | 11 | 4
Not completed — Decision of Participant | 0 | 1 | 3
Not completed — Adverse Event | 0 | 9 | 1
Not completed — Other Miscellaneous Reasons | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who had ocular inserts placed in their eyes.
Groups:
- Total: Total of all reporting groups
Arm/Group | 13 mg Bimatoprost Ocular Insert | Timolol 0.5% + Placebo Ocular Insert | Total
Number analyzed (Participants) | 64 | 66 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (10.1) | 66.3 (8.5) | 65.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 44 | 77
  Male | 31 | 22 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intra-Ocular Pressure (IOP) at Week 2
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP measurements were taken at 8 am (time (T)=0 hour), 10 am (T=2 hour), and 4 pm (T=8 hour) at Week 2. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0) to Week 2
Population: Participants from the Full Analysis Set (FAS), all randomized participants who had ocular inserts placed in their eye and who had at least 1 on-treatment study visit completed, with data available for analysis at the given time-point.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | 13 mg Bimatoprost Ocular Insert | Timolol 0.5% + Placebo Ocular Insert
Number analyzed (Participants) | 63 | 64
mm Hg
  Baseline (T=0 hour) | 24.99 (0.29) | 25.34 (0.29)
  Baseline (T=2 hour) | 23.65 (0.31) | 23.75 (0.28)
  Baseline (T=8 hour) | 22.95 (0.29) | 23.16 (0.29)
  Change from Baseline to Week 2 (T=0 hour): number analyzed (Participants) | 63 | 63
  Change from Baseline to Week 2 (T=0 hour) | -6.40 (0.41) | -6.30 (0.41)
  Change from Baseline to Week 2 (T=2 hour): number analyzed (Participants) | 63 | 63
  Change from Baseline to Week 2 (T=2 hour) | -5.20 (0.34) | -5.59 (0.41)
  Change from Baseline to Week 2 (T=8 hour): number analyzed (Participants) | 62 | 63
  Change from Baseline to Week 2 (T=8 hour) | -4.21 (0.35) | -4.96 (0.37)

2. Primary Outcome: Change From Baseline in Intra-Ocular Pressure (IOP) at Week 6
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP measurements were taken at 8 am (T=0 hour), 10 am (T=2 hour), and 4 pm (T=8 hour) at Week 6. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0) to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | 13 mg Bimatoprost Ocular Insert | Timolol 0.5% + Placebo Ocular Insert
Number analyzed (Participants) | 63 | 64
mm Hg
  Baseline (T=0 hour) | 24.99 (0.29) | 25.34 (0.29)
  Baseline (T=2 hour) | 23.65 (0.31) | 23.75 (0.28)
  Baseline (T=8 hour) | 22.95 (0.29) | 23.16 (0.29)
  Change from Baseline to Week 6 (T=0 hour): number analyzed (Participants) | 60 | 64
  Change from Baseline to Week 6 (T=0 hour) | -5.47 (0.40) | -6.41 (0.41)
  Change from Baseline to Week 6 (T=2 hour): number analyzed (Participants) | 60 | 64
  Change from Baseline to Week 6 (T=2 hour) | -4.70 (0.31) | -5.40 (0.39)
  Change from Baseline to Week 6 (T=8 hour): number analyzed (Participants) | 60 | 63
  Change from Baseline to Week 6 (T=8 hour) | -3.78 (0.34) | -4.42 (0.39)

3. Primary Outcome: Change From Baseline in Intra-Ocular Pressure (IOP) at Week 12
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP measurements were taken at 8 am (T=0 hour), 10 am (T=2 hour), and 4 pm (T=8 hour) at Week 12. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0) to Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | 13 mg Bimatoprost Ocular Insert | Timolol 0.5% + Placebo Ocular Insert
Number analyzed (Participants) | 63 | 64
mm Hg
  Baseline (T=0 hour) | 24.99 (0.29) | 25.34 (0.29)
  Baseline (T=2 hour) | 23.65 (0.31) | 23.75 (0.28)
  Baseline (T=8 hour) | 22.95 (0.29) | 23.16 (0.29)
  Change from Baseline to Week 12 (T=0 hour): number analyzed (Participants) | 57 | 63
  Change from Baseline to Week 12 (T=0 hour) | -5.26 (0.47) | -6.31 (0.43)
  Change from Baseline to Week 12 (T=2 hour): number analyzed (Participants) | 57 | 63
  Change from Baseline to Week 12 (T=2 hour) | -4.26 (0.44) | -5.60 (0.43)
  Change from Baseline to Week 12 (T=8 hour): number analyzed (Participants) | 57 | 63
  Change from Baseline to Week 12 (T=8 hour) | -3.99 (0.33) | -5.19 (0.35)

4. Secondary Outcome: Change From Baseline in IOP at Month 4
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP measurements were taken at 8 am (T=0 hour), 10 am (T=2 hour), and 4 pm (T=8 hour) at Month 4. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 1) to Month 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | 13 mg Bimatoprost Ocular Insert | Timolol 0.5% + Placebo Ocular Insert
Number analyzed (Participants) | 63 | 64
mm Hg
  Baseline (T=0 hour) | 24.99 (0.29) | 25.34 (0.29)
  Baseline (T=2 hour) | 23.65 (0.31) | 23.75 (0.28)
  Baseline (T=8 hour) | 22.95 (0.29) | 23.16 (0.29)
  Change from Baseline to Month 4 (T=0 hour): number analyzed (Participants) | 54 | 63
  Change from Baseline to Month 4 (T=0 hour) | -5.14 (0.43) | -6.29 (0.40)
  Change from Baseline to Month 4 (T=2 hour): number analyzed (Participants) | 54 | 63
  Change from Baseline to Month 4 (T=2 hour) | -4.37 (0.38) | -5.26 (0.41)
  Change from Baseline to Month 4 (T=8 hour): number analyzed (Participants) | 54 | 63
  Change from Baseline to Month 4 (T=8 hour) | -3.84 (0.34) | -5.11 (0.36)

5. Secondary Outcome: Change From Baseline in IOP at Month 5
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP measurements were taken at 8 am (T=0 hour), 10 am (T=2 hour), and 4 pm (T=8 hour) at Month 5. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0) to Month 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | 13 mg Bimatoprost Ocular Insert | Timolol 0.5% + Placebo Ocular Insert
Number analyzed (Participants) | 63 | 64
mm Hg
  Baseline (T=0 hour) | 24.99 (0.29) | 25.34 (0.29)
  Baseline (T= 2 hour) | 23.65 (0.31) | 23.75 (0.28)
  Baseline (T=8 hour) | 22.95 (0.29) | 23.16 (0.29)
  Change from Baseline to Month 5 (T=0 hour): number analyzed (Participants) | 53 | 63
  Change from Baseline to Month 5 (T=0 hour) | -4.28 (0.36) | -6.35 (0.41)
  Change from Baseline to Month 5 (T=2 hour): number analyzed (Participants) | 53 | 63
  Change from Baseline to Month 5 (T=2 hour) | -3.87 (0.39) | -5.45 (0.43)
  Change from Baseline to Month 5 (T=8 hour): number analyzed (Participants) | 53 | 63
  Change from Baseline to Month 5 (T=8 hour) | -3.21 (0.34) | -4.47 (0.38)

6. Secondary Outcome: Change From Baseline in IOP at Month 6
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP measurements were taken at 8 am (T=0 hour), 10 am (T=2 hour), and 4 pm (T=8 hour) at Month 6. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0) to Month 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | 13 mg Bimatoprost Ocular Insert | Timolol 0.5% + Placebo Ocular Insert
Number analyzed (Participants) | 63 | 64
mm Hg
  Baseline (T=0 hour) | 24.99 (0.29) | 25.34 (0.29)
  Baseline (T=2 hour) | 23.65 (0.31) | 23.75 (0.28)
  Baseline (T=8 hour) | 22.95 (0.29) | 23.16 (0.29)
  Change from Baseline to Month 6 (T=0 hour): number analyzed (Participants) | 53 | 62
  Change from Baseline to Month 6 (T=0 hour) | -4.58 (0.39) | -5.97 (0.42)
  Change from Baseline to Month 6 (T=2 hour): number analyzed (Participants) | 53 | 62
  Change from Baseline to Month 6 (T=2 hour) | -3.87 (0.42) | -5.20 (0.41)
  Change from Baseline to Month 6 (T=8 hour): number analyzed (Participants) | 53 | 62
  Change from Baseline to Month 6 (T=8 hour) | -3.25 (0.32) | -4.24 (0.37)

ADVERSE EVENTS:
Time Frame: Randomization (Day 0) to the end of study (Up to 6 Months)
Arm/Group | 13 mg Bimatoprost Ocular Insert | Timolol 0.5% + Placebo Ocular Insert
Serious Adverse Events (participants affected / at risk) | 1/64 | 2/66
Other Adverse Events (participants affected / at risk) | 20/64 | 14/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13 mg Bimatoprost Ocular Insert (N=64) | Timolol 0.5% + Placebo Ocular Insert (N=66)
Hypertension (Vascular disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 13 mg Bimatoprost Ocular Insert (N=64) | Timolol 0.5% + Placebo Ocular Insert (N=66)
Eye discharge (Eye disorders) | 7 | 7
Conjunctival hyperaemia (Eye disorders) | 9 | 2
Punctate keratitis (Eye disorders) | 5 | 4
Eye pruritus (Eye disorders) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No presentation or publication of Institution's data relating to the Trial may occur until after the Trial has been completed at all sites. If Investigator desires to present or publish, investigator must submit any and all manuscripts, posters, abstracts, or other intended publications (hereinafter collectively referred to as "manuscripts") to Sponsor at least sixty (60) days prior to the actual submission of such manuscript(s) for publication.